CLINICAL TRIAL: NCT05750355
Title: A Single-dose-oral, Ascending-Dose, Single-Center,Randomized, Double-Blind, Placebo-Parallel-controlled Study for the Evaluation of the Effect of TPN171H Tablets on the QT/QTc Intervals in Adult Healthy Subjects
Brief Title: Evaluate the Effect of TPN171H on the QT/QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPN171H-11
Record Dates: First submitted 2022-11-06; First posted 2023-03-01 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Healthy Subjects
Keywords: TPN171H tablets; QT/QTc Intervals
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPN171H (Experimental): Subjects will receive TPN171H orally for single dose
  Interventions: Drug: TPN171H 10 mg Group; Drug: TPN171H 30 mg Group; Drug: TPN171H 40 mg Group; Drug: TPN171H 50 mg Group
- Placebo (Placebo Comparator): Subjects will receive Placebo orally for single dose
  Interventions: Drug: TPN171H 10 mg Group; Drug: TPN171H 30 mg Group; Drug: TPN171H 40 mg Group; Drug: TPN171H 50 mg Group

INTERVENTIONS:
Drug: TPN171H 10 mg Group — 6 subjects will receive TPN171H 10 mg, orally; 2 subjects will receive placebo, orally.
  Other Names: TPN171H 10 mg
Drug: TPN171H 30 mg Group — 6 subjects will receive TPN171H 30 mg, orally; 2 subjects will receive placebo, orally.
  Other Names: TPN171H 30 mg
Drug: TPN171H 40 mg Group — 6 subjects will receive TPN171H 40 mg, orally; 2 subjects will receive placebo, orally.
  Other Names: TPN171H 40 mg
Drug: TPN171H 50 mg Group — 6 subjects will receive TPN171H 50 mg, orally; 2 subjects will receive placebo, orally.
  Other Names: TPN171H 50 mg

SUMMARY:
This is a single-dose orally administered, dose-escalation, single-center, randomized, double-blind, placebo-parallel controlled clinical study evaluating the effect of TPN171H tablets on QT/QTc interval in healthy subjects.The main objective was to evaluate the effect of TPN171H tablets on QT/QTc interval in healthy Chinese subjects after a single oral administration.

DETAILED DESCRIPTION:
This trial was a single-center, randomized, double-blind, placebo parallel controlled trial of TPN171H tablets with single oral administration, dose escalation, in healthy Chinese subjects.

This trial plans to set up 4 dose groups, and a total of 32 healthy adult subjects are expected to be enrolled. All subjects will receive a single oral dose under fasting state, and complete 3 days of PK blood sampling, 12-lead ECG examination and other safety checks. The trial was sequential according to the principle of dose escalation, that is, the next dose group was tested on the premise that the safety and tolerability of the previous group were good.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years old, both male and female;
2. Weight: male ≥ 50 kg, female ≥ 45 kg, 19 kg/m2 ≤ BMI ≤26 kg/m2
3. Three 12-lead ECG examinations (the average of three measurements will be used to determine eligibility), QTcF≤450 ms, PR interval ≤200 ms, and QRS duration <120 ms;
4. Reliable contraceptive measures will be taken from the signing of the informed consent to 3 months after the medication, and there is no plan to donate sperm or eggs. The specific contraceptive measures are detailed in the appendix.
5. Able to understand the procedures and methods of this trial, willing to strictly abide by the clinical trial protocol to complete this trial, and voluntarily sign the informed consent.

Exclusion Criteria:

1. Known allergic history to the investigational drug and any of its components or related preparations;
2. People with allergic diseases, food allergies or allergic constitutions;
3. have a history of risk factors for torsdos de pointes, or have a family history of short QT syndrome, long QT syndrome, unexplained sudden death in young adulthood (≤40 years old), drowning or sudden infant death syndrome in first-degree relatives (i.e., biological parents, siblings or children);
4. Previous history of hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia;
5. Those who have definite diseases of the central nervous system, cardiovascular system, digestive system (including those with moderate or severe fatty liver on B-ultrasound examination), respiratory system, urinary system, blood system, and metabolic disorders that require medical intervention or other diseases that are not suitable for clinical trials (such as psychiatric history, etc.);
6. Patients with blurred vision or history of ophthalmology (such as abnormal color vision, retinitis pigmentosa, macular degeneration);
7. Patients with a history of postural hypotension;
8. Patients with a history of acute respiratory infection or acute illness within 14 days before screening;
9. Those who had donated blood or lost ≥400 mL of blood within 3 months before screening;
10. Use of any drugs that inhibit or induce liver metabolism of drugs (such as: inducers - barbiturates, carbazepine, phenytoin, glucocorticoids, omeprazole; Inhibitors -SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazole, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines);
11. Those who have taken any prescription drugs, non-prescription drugs, health care products, vitamins and Chinese herbal medicines within 14 days before screening;
12. Consuming grapefruit, grapefruit, pitaya, mango and other fruits or related products that affect metabolic enzymes within 7 days before screening;
13. Intake of caffeine-rich or xanthine-rich beverages or foods (such as coffee, strong tea, chocolate, cola, etc.) within 48 h before screening;
14. Those who participated in other drug clinical trials within 3 months before screening;
15. Current or former drug users or alcohol addicts, current or former alcoholics (drinking more than 14 standard units per week). 1 standard unit containing 14g of alcohol (e.g. 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or a positive breath test for alcohol;
16. Those who smoked more than 10 cigarettes per day in the previous 3 months were screened;
17. Physical examination, abnormal vital signs (ear temperature >37.5℃, respiratory rate >20 beats/minute, pulse rate >100 beats/minute, systolic blood pressure ≥140 mmHg or <90 mmHg, diastolic blood pressure ≥90 mmHg or <50 mmHg), abnormal and clinically significant laboratory results, and those who have an impact on the evaluation of this trial;
18. Laboratory tests showed that serum potassium, magnesium and calcium were beyond the normal range and the abnormalities were judged by the researchers to be clinically significant;
19. Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, syphilis antibody (TPPA) or human immunodeficiency virus (HIV) antibody positive;
20. Abnormal chest X-ray (anteroposterior and lateral view) or lung CT results with clinical significance;
21. Women with positive blood pregnancy test (applicable to women) or lactating women;
22. Those who have other factors that the investigator considers unsuitable for participation in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
QT Interval Corrected Using Fridericia's Formula | From Day 1 to Day3
  Model-guided placebo-corrected change in QTcF from baseline (ΔΔQTcF)

SECONDARY OUTCOMES:
QT Interval | From Day 1 to Day3
  Change in QT interval from baseline
Corrected QT interval | From Day 1 to Day3
  Change in QTc interval from baseline
PR interval | From Day 1 to Day3
  Change in PR interval from baseline
RR interval | From Day 1 to Day3
  Change in RR interval from baseline
QRS duration | From Day 1 to Day3
  Change in QRS duration limit interval from baseline
Heart rate | From Day 1 to Day3
  Change in HR from baseline
T-wave | From Day 1 to Day3
  Whether the T-wave shape is abnormal
U-wave | From Day 1 to Day3
  Whether the U-wave shape is abnormal
Number of participants with arrhythmic | From Day 1 to Day3
  Number of participants with arrhythmic, arrhythmic includes Atrial fibrillation, atrial flutter, atrioventricular block, ST segment changes, etc
Tmax | From Day 1 to Day3
  time to peak
Cmax | From Day 1 to Day3
  maximum concentration
plasma half-life（T1/2） | From Day 1 to Day3
  Elimination half life
Area under concentration-time curve (AUC0-t) | From Day 1 to Day3
  Area under concentration-time curve (AUC0-t)
Incidence of adverse events | From Day 1 to Day3
  Incidence of adverse events
Severity of adverse events | From Day 1 to Day3
  Severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China